CLINICAL TRIAL: NCT07340073
Title: Coordinated Reset Deep Brain Stimulation for Parkinson's Disease
Acronym: CR DBS PD
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NEUR-2025-34279
Record Dates: First submitted 2025-11-13; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Parkinson's Disease (PD); Deep Brain Stimulation
Keywords: Deep Brain Simulation; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- CR-DBS (Active Comparator): Randomized to either T-DBS occurring first or CR-DBS occurring first (50/50 chance of being assigned to either, but will be assessing both)
  Interventions: Device: DBS
- T-DBS (Active Comparator): Randomized to either T-DBS occurring first or CR-DBS occurring first (50/50 chance of being assigned to either, but will be assessing both)
  Interventions: Device: DBS

INTERVENTIONS:
Device: DBS — Deep Brain Stimulation

SUMMARY:
Deep brain stimulation (DBS) is a surgical implant procedure for the treatment of Parkinson's Disease (PD) utilizing medical devices approved by the FDA. A novel approach to current DBS approaches is called "Coordinated Reset" DBS (CR-DBS) which uses different patterns of stimulation at lower currents and can address the limitations of traditional DBS (T-DBS) that uses continuous high amplitude and high frequency stimulation. This study will evaluate the safety and short-term efficacy of CR-DBS in PD. The results from this study will significantly advance the development of CR-DBS for the treatment of PD. Findings in this study will also provide the rationale for further development of this novel DBS approach for other neurological and psychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Idiopathic Parkinson's Disease
* Minimum age of 21 years old
* Will be or has been implanted with the Boston Scientific Vercise Genus Rechargeable DBS system

Exclusion Criteria:

* History of musculoskeletal disorders that affect movement of the limbs/gait
* Other significant neurological disorder
* Significant psychiatric disorder
* History of dementia or cognitive impairment that precludes them from getting DBS surgery or per study staff judgment, MacCAT-CR assessment does not deduce that the participant has capacity to consent
* Other significant medical disorder that could impede study participation
* Pregnant women

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2031-01-01 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
Movement Disorder Society-Unified Parkinson's Disease Rating Scale Part III | Through participant study completion, an average of two months
  The MDS-UPDRS is a standard rating scale for PD that has been widely used in clinical settings and PD research. It utilizes a 4-subscale structure and 5-point (Normal = 0 to Severe = 4) severity scale. Part III of the Scale assesses the motor signs of PD through 18 items, with a maximum possible score of 72.

SECONDARY OUTCOMES:
Frequency and Severity of Bradykinesia, Dyskinesia, Tremor, Sleep Quality and Fragmentation Scores Measured via KinetiGraph. | Through participant study completion, an average of two months
  The KinetiGraph PKG system consists of a small watch-device worn on the wrist for collecting data over a period of several days and provides a report that shows how motor symptoms and complications of PD such as bradykinesia, tremor and dyskinesias vary throughout the day. The watch will be worn on the patient's most affected side (indicated by each patient's MDS-UPDRS III scores for two body sides).
Amplitude Decrement via Rapid Alternating Movements (RAMs) | Through participant study completion, an average of two months
  This task assesses hypokinesia and the sequence effect (deterioration of movement amplitude over time). Pronation-supination movements will be performed using a forearm manipulandum. Movement will be visually guided and acoustically paced. Four 60-second trials will be completed each side (right and left arms), with each trial including 4 transitions in movement rate (1.0 or 1.75 Hz). Delsys inertial measurement units (IMUs) will also be used during this task to measure EMG and kinematic data.
Forearm Rigidity | Through participant study completion, an average of two months
  Forearm rigidity will be assessed using a custom-built robotic manipulandum which provides reliable and objective measures of resistance to imposed motion. The device passively imposes sinusoidal movements of the forearm about the pronation-supination axis through a ± 40° range of motion at 1.5 Hz while measuring the angular displacement and resistive torque required to move the limb. Trials will be collected separately for the right and left arms, with or without an activation maneuver (tapping the contralateral hand on the leg), a technique that is used clinically to elicit or enhance rigidity. Delsys inertial measurement units (IMUs) will be used to measure the EMG activities of biceps brachii and pronator teres muscles, as secondary measurements during the task.
Cognitive Measurements (TMT-B) | Through participant study completion, an average of two months
  Trail Making Task-B will evaluate visual scanning, sequencing, cognitive flexibility and processing speed will be completed.
Verbal Fluency Measurement (DKEFS) | Through participant study completion, an average of two months
  DKEFS Verbal Fluency Task will evaluate verbal fluency.
Working Memory Assessment via N-Back Task | Through participant study completion, an average of two months
  Quantitative assessment of accuracy and reaction time as a function of working memory load.
Dyskinesia Assessment via Rush Dyskinesia Rating Scale (RDRS) | Through participant study completion, an average of two months
  RDRS will assess the severity of overall dyskinesias during activities of daily living. A severity rating score of 4 indicates violent dyskinesia and 0 indicates an absence of dyskinesia. This scale can also distinguish chorea from dystonia (the two major types of dyskinesias in PD) and identify the single most disabling form of dyskinesia.
Frequency of participants with adverse events as assessed by CTCAE v6.0 | Through participant study completion, an average of two months
  Frequency [between and within] participants with treatment-related adverse events as assessed by CTCAE v6.0. This is a qualitative collection of information via participant report or clinical observation, but will be input as quantitative (e.g., a headache can be classified as "1-Mild, 2-Moderate, and 3-Severe).
Step Length ("Steady-State Gait") | Through participant study completion, an average of two months
  In this gait task, spatial and temporal gait metrics will be obtained using wearable inertial measurement units (IMUs) on the feet, wrists, lumbar, and sternum. Patients will walk for ~1 minute, back and forth along a ~12m walkway, followed by ~1 minute of rest (repeated 5x)
Gait Speed ("Steady-State Gait") | Through participant study completion, an average of two months
  In this gait task, spatial and temporal gait metrics will be obtained using wearable inertial measurement units (IMUs) on the feet, wrists, lumbar, and sternum. Patients will walk for ~1 minute, back and forth along a ~12m walkway, followed by ~1 minute of rest (repeated 5x)
Cadence ("Steady-State Gait") | Through participant study completion, an average of two months
  In this gait task, spatial and temporal gait metrics will be obtained using wearable inertial measurement units (IMUs) on the feet, wrists, lumbar, and sternum. Patients will walk for ~1 minute, back and forth along a ~12m walkway, followed by ~1 minute of rest (repeated 5x)
Step Variability ("Steady-State Gait") | Through participant study completion, an average of two months
  In this gait task, spatial and temporal gait metrics will be obtained using wearable inertial measurement units (IMUs) on the feet, wrists, lumbar, and sternum. Patients will walk for ~1 minute, back and forth along a ~12m walkway, followed by ~1 minute of rest (repeated 5x)
Step Asymmetry ("Steady-State Gait") | Through participant study completion, an average of two months
  In this gait task, spatial and temporal gait metrics will be obtained using wearable inertial measurement units (IMUs) on the feet, wrists, lumbar, and sternum. Patients will walk for ~1 minute, back and forth along a ~12m walkway, followed by ~1 minute of rest (repeated 5x)
Swing Time Variability ("Steady-State Gait") | Through participant study completion, an average of two months
  In this gait task, spatial and temporal gait metrics will be obtained using wearable inertial measurement units (IMUs) on the feet, wrists, lumbar, and sternum. Patients will walk for ~1 minute, back and forth along a ~12m walkway, followed by ~1 minute of rest (repeated 5x)
Frequency of Freezing of Gait ("Steady-State Gait") | Through participant study completion, an average of two months
  In this gait task, spatial and temporal gait metrics will be obtained using wearable inertial measurement units (IMUs) on the feet, wrists, lumbar, and sternum. Patients will walk for ~1 minute, back and forth along a ~12m walkway, followed by ~1 minute of rest (repeated 5x)
Duration of Freezing of Gait ("Steady-State Gait") | Through participant study completion, an average of two months
  In this gait task, spatial and temporal gait metrics will be obtained using wearable inertial measurement units (IMUs) on the feet, wrists, lumbar, and sternum. Patients will walk for ~1 minute, back and forth along a ~12m walkway, followed by ~1 minute of rest (repeated 5x)
Difference in Step Length (w/ and w/o 1-Back; "Dual-Task Effect on Gait") | Through participant study completion, an average of two months
  The dual-task effect on gait will be assessed by repeating the gait task; spatial and temporal gait metrics will be obtained using wearable inertial measurement units (IMUs) on the feet, wrists, lumbar, and sternum. Patients will walk for ~1 minute, back and forth along a ~12m walkway, followed by ~1 minute of rest while the patient performs a 1-back cognitive task.
Difference in Gait Speed (w/ and w/o 1-Back; "Dual-Task Effect on Gait") | Through participant study completion, an average of two months
  The dual-task effect on gait will be assessed by repeating the gait task; spatial and temporal gait metrics will be obtained using wearable inertial measurement units (IMUs) on the feet, wrists, lumbar, and sternum. Patients will walk for ~1 minute, back and forth along a ~12m walkway, followed by ~1 minute of rest while the patient performs a 1-back cognitive task.
Difference in Cadence (w/ and w/o 1-Back; "Dual-Task Effect on Gait") | Through participant study completion, an average of two months
  The dual-task effect on gait will be assessed by repeating the gait task; spatial and temporal gait metrics will be obtained using wearable inertial measurement units (IMUs) on the feet, wrists, lumbar, and sternum. Patients will walk for ~1 minute, back and forth along a ~12m walkway, followed by ~1 minute of rest while the patient performs a 1-back cognitive task.
Difference in Step Variability (w/ and w/o 1-Back; "Dual-Task Effect on Gait") | Through participant study completion, an average of two months
  The dual-task effect on gait will be assessed by repeating the gait task; spatial and temporal gait metrics will be obtained using wearable inertial measurement units (IMUs) on the feet, wrists, lumbar, and sternum. Patients will walk for ~1 minute, back and forth along a ~12m walkway, followed by ~1 minute of rest while the patient performs a 1-back cognitive task.
Difference in Step Asymmetry (w/ and w/o 1-Back; "Dual-Task Effect on Gait") | Through participant study completion, an average of two months
  The dual-task effect on gait will be assessed by repeating the gait task; spatial and temporal gait metrics will be obtained using wearable inertial measurement units (IMUs) on the feet, wrists, lumbar, and sternum. Patients will walk for ~1 minute, back and forth along a ~12m walkway, followed by ~1 minute of rest while the patient performs a 1-back cognitive task.
Difference in Swing Time Variability (w/ and w/o 1-Back; "Dual-Task Effect on Gait") | Through participant study completion, an average of two months
  The dual-task effect on gait will be assessed by repeating the gait task; spatial and temporal gait metrics will be obtained using wearable inertial measurement units (IMUs) on the feet, wrists, lumbar, and sternum. Patients will walk for ~1 minute, back and forth along a ~12m walkway, followed by ~1 minute of rest while the patient performs a 1-back cognitive task.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wang, PhD, Principal Investigator — University of Minnesota

IPD SHARING:
Plan to Share IPD: No